CLINICAL TRIAL: NCT05963828
Title: COmprehensive Management of High-risk PopuLatIon of Stroke bAsed oN soCial nEtwork: a Multicenter, Parallel and Randomized Controlled sTudy
Brief Title: Comprehensive Management of High-risk PopuLatIon of Stroke Based on Social Network
Acronym: COMPLIANCE-MT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Changhai Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: COMPLIANCE-MT
Record Dates: First submitted 2023-04-14; First posted 2023-07-27 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Stroke; Cerebrovascular Disorders; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Vascular Diseases; Cardiovascular Diseases
Keywords: Stroke; Management; Social Networks
MeSH Terms: conditions — Stroke; Cerebrovascular Disorders; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Vascular Diseases; Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard group (Other): Patients are managed according to the routine methods after enrollment.
  Interventions: Behavioral: Routine post-hospital follow-up management
- Experimental group (Experimental): Patients are managed by the social network platform.
  Interventions: Behavioral: Post-hospital management based on WeChat applet

INTERVENTIONS:
Behavioral: Post-hospital management based on WeChat applet — The brain and heart health manager uses the exclusive QR code in the WeChat applet to receive and manage patients. Patients can register and use the WeChat applet by scanning the QR code. The functions of WeChat applet include making medication plan for patients, daily medication reminder, targeted health education, health index monitoring, online consultation and so on.
  Arms: Experimental group
Behavioral: Routine post-hospital follow-up management — The brain and mental health managers routinely followed up the patients in the standard group for 1, 3, 6 and 12 months by telephone or outpatient follow-up, the main content of which was to inquire about the medication of patients and the management of stroke risk factors. Targeted health education was carried out according to the risk factors of patients.
  Arms: Standard group

SUMMARY:
The purpose of this study is to evaluate the effectiveness of social network in improving drug compliance and risk factors control rate of stroke high-risk population after discharge.

DETAILED DESCRIPTION:
Stroke is the leading cause of death among residents in China, with the characteristics of high morbidity, high mortality, high disability rate, high recurrence rate and so on, which brings huge economic burden to the patients' families and society. Strengthening the comprehensive management of the high-risk population of stroke, improving the medication compliance of patients and the control rate of stroke risk factors play a key role in reducing stroke recurrence.

This study is a multicenter, prospective, randomized, single-blind study, which aims to use the tool of WeChat Mini Programs to realize the post-hospital follow-up management of the high-risk population of stroke. The follow-up time is 12 months. The main measurement result was the change of patients' medication compliance after comprehensive management.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* High-risk population of stroke for hospitalization
* Modified Rankin Scale score≤ 2
* Patients or primary caregiver have smart phone and wechat accounts
* Patients take at least one drug for a long time (antihypertensive, hypoglycemic, lipid-lowering, anticoagulant, antiplatelet drugs)
* Written informed consent

Exclusion Criteria:

* Patients and their families are unable to operate smartphones
* Having other diseases that interfere with clinical follow-up assessment (such as cancer, dementia, severe mental illness, etc.)
* Life expectancy is less than 12 months
* Patients living in the absence of network conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 720 (Estimated)
Dates: Start 2023-07-18 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Patient's medication adherence to five evidence-based secondary prevention drugs for stroke at 12 months after discharge | 12 months after discharge
  Compliance is defined when patients take all evidence-based secondary preventive drugs (antihypertensive, hypoglycemic, lipid-regulating, anticoagulant and antiplatelet drugs) for more than 24 days in 12 months after discharge, that is, the drug taking rate is > 80% (> 24/30 days). If the patient adjusts the drug or stops taking the drug by himself, it will be regarded as "non-compliance". If the patient stops taking the drug according to the doctor's advice, it will be regarded as compliance. If the drug is adjusted according to the doctor's advice, it is necessary to continue to ask about the number of days of taking the drug in the past month. If the number of days of taking the drug exceeds 24 days, it will be regarded as compliance.

SECONDARY OUTCOMES:
The rate of good compliance with stroke prevention drugs among patients 1 month, 3 months, 6 months and 12 months after discharge | 1 month, 3 months，6 months and 12 months after discharge.
  Measured by Morisky Medication Adherence Scale 8 item; Morisky Medication Adherence Scale 8 item
The attainment rate of stroke risk factors (blood glucose, blood pressure, blood lipid, BMI, waist circumference, hip circumference, smoking) at 1 month, 3 months, 6 months and 12 months after discharge. | 1 month, 3 months, 6 months and 12 months after discharge
  The method of measurement is as follows:
  Blood lipids: fasting blood sampling measurement Blood glucose: fasting fingertip blood glucose Blood pressure: using a sphygmomanometer to measure BMI: weight (kg) / height (m) ^ 2 Waist circumference, Hip circumference, Smoking: Patient self-report
Knowledge of stroke | 1 month, 3 months, 6 months and 12 months after discharge
  Measured by The Knowledge questionnaire on prevention and treatment of stroke
Personal motivation | 1 month, 3 months, 6 months and 12 months after discharge
  Measured by The Stroke Attitude Questionnaire
Stroke health behavior improvement | 1 month, 3 months, 6 months and 12 months after discharge
  Measured by The Stroke Prevention Health Behavior Scale
Social motivation | 1 month, 3 months, 6 months and 12 months after discharge
  Measured by Perceived Social Support Scale
Health-related quality of life | 1 month, 3 months, 6 months and 12 months after discharge
  Measured by The 5-level EQ-5D
Incidence of anxiety | 1 month, 3 months, 6 months and 12 months after discharge
  Measured by Generalized Anxiety Disorder-7
Incidence of depression | 1 month, 3 months, 6 months and 12 months after discharge
  Measured by Patient Health Questionnaire-9
Self efficacy | 1 month, 3 months, 6 months and 12 months after discharge
  Measured by Chronic Disease Self-Efficacy Scale
Incidence of major cardiovascular events including stroke, acute coronary syndrome, and vascular death | 1 month, 3 months, 6 months and 12 months after discharge
  Stroke: cerebral blood supply disorder caused by acute (focal) neurological syndrome, there is ischemic or hemorrhagic lesion in the corresponding area on brain imaging, or clinical evidence shows negative ischemic lesion on imaging, and the symptoms last longer than 24 hours.
  Acute coronary syndrome: ①typical clinical symptoms (such as chest pain, heart failure, etc.) accompanied by typical electrocardiogram (ECG) abnormalities; ② typical clinical symptoms with troponin elevated more than 2 times the upper limit of normal;③ or Non-specific symptoms with elevated troponin more than 2 times the upper limit of normal; ④Asymptomatic myocardial infarction diagnosed by follow-up ECG compared with baseline ECG combined with corresponding results of echocardiography or coronary angiography.
  Vascular death: including death within 30 days after stroke, death within 7 days after acute coronary syndrome, non-cerebral hemorrhage or necrotic death after peripheral artery occlusion or

CONTACTS AND LOCATIONS:
Overall Officials: Zhang lingjuan, Study Director — Changhai Hospital
Locations (1):
- Changhai Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No